CLINICAL TRIAL: NCT00598104
Title: A Randomized, Double-blinded, Placebo Controlled, Parallel Group, Multi-center Study to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of Intravenous Doses of QAX576 in Moderate Persistent Allergic Asthmatics Following Inhaled Corticosteroid Withdrawal
Brief Title: Safety and Efficacy of QAX576 in Adults With Moderate Persistent Allergic Asthma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the lack of enrolment and complexity of design, this study in asthma was terminated. No subjects have been dosed for this study.
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAX576A2103
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: Asthma, interleukin-13
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: QAX576
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAX576
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study will evaluate the safety and efficacy of QAX576 against asthma attacks in adults with moderate persistent allergic asthma

ELIGIBILITY:
Inclusion Criteria:

* History of asthma attacks
* Taking inhaled corticosteroids
* Non-smoking

Exclusion Criteria:

* Women of child-bearing potential
* History of respiratory disease other than asthma
* History of severe allergy to food or drugs
* Previous use of monoclonal antibodies
* Very low or high body weight

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
- Forced expiratory volume in 1 second (FEV1)at baseline and until study completion - Levels of eosinophils in sputum | Throughout the study

SECONDARY OUTCOMES:
- Three doses of QAX576 on time to treatment failure, plasma IL-13 levels and immunogenicity in asthmatics - Sputum biomarkers | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigative site